CLINICAL TRIAL: NCT03088007
Title: Importance of Multidimensional Assessments in Accompanying Schooling of Children With Mild to Moderate Intellectual Disability.
Acronym: EVAL'ID
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0257
Record Dates: First submitted 2017-03-10; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Disability, Intellectual
Keywords: Intellectual Deficiency; cognitive, adaptive; behavioral and academic profile; regular and special schools
MeSH Terms: conditions — Intellectual Disability; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IME attending ID children: Children with mild to moderate Intellectual Deficiency attending school at IME (Instituts Médico-Educatifs, which are special schools mandated to accommodate children and young people with Intellectual Disability at any level of disability).
  Interventions: Other: Cognitive, adaptive, behavioral and academic assessment
- ULIS attending ID children: Children with mild to moderate Intellectual Deficiency attending school at ULIS (Unités Localisées pour l'Inclusion Scolaire, which enables disabled children to attend regular schools)
  Interventions: Other: Cognitive, adaptive, behavioral and academic assessment

INTERVENTIONS:
Other: Cognitive, adaptive, behavioral and academic assessment — Cognitive, adaptive, behavioral and academic assessment will be performed if not available in the records, using WISC-IV, VABS, GECEN and an academic skills rating form.

SUMMARY:
The EVAL'ID study aims to demonstrate the value of a multidimensional assessment in accompanying schooling of children with Intellectual Disability. The study will be performed in the Rhône department (France) in children aged from 5 to 13 years with mild to moderate Intellectual Disability , and attending school either at ULIS (Unités Localisées pour l'Inclusion Scolaire, which enables disabled children to attend regular schools), or IME (Instituts Médico-Educatifs, which are special schools mandated to accommodate children and young people with Intellectual Disability at any level of disability). A multidimensional assessment encompasses the assessment of academic, cognitive, behavioral and adaptive skills of the children, with validated and reliable neuropsychological batteries, called ID Kit (Intellectual Deficiency assessment Kit), which includes the following scales : the Wechsler Intelligence Scale for Children 4th edition (WISC-IV), the Vineland Adaptive Behavioral Scale II, the GECEN rating form (Grille d'Evaluation Comportementale pour Enfants Nisonger, which is the French translation of the Nisonger Child Behavior Rating Form), and an academic skills rating form (GEVA-SCO). A comparison of the children neuropsychological profiles according to the type of school they attend, will be perform.

The project consists of three phases:

* Stage 1: Collection of information from each child records at MDPH (Departmental Administration for Disabled Persons), IME, ULIS schools, including the assessments that were performed, and from a survey of both caregivers and parents regarding their respective perception and knowledge of the child's disability
* Stage 2: All the children who were not previously assessed with the ID kit will be further evaluated using these tests. The results of these assessments will be shared with parents and caregivers.
* Stage 3: A survey regarding the perception and knowledge of the child's disability will be carried out again among caregivers and parents.

ELIGIBILITY:
Inclusion Criteria:

* Age : > 5 and <13 years
* With mild to moderate intellectual deficiency
* attending school either at ULIS or IME in the Rhône department.

Exclusion Criteria:

* No insurance coverage
* No parents agreement

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged from 5 to 13 years with mild to moderate Intellectual Disability , and attending school either at ULIS (Unités Localisées pour l'Inclusion Scolaire, which enables disabled children to attend regular schools), or IME (Instituts Médico-Educatifs, which are special schools mandated to accommodate children and young people with Intellectual Disability at any level of disability), within the Rhône department, France.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Presence of the ID assessment kit results in the records | within one year before the latest child orientation decision
  The primary outcome measure consists of the presence of the results of the neuropsychological tests included in the ID assessment kit: WISC-IV (IQ), Vineland Adaptive Behavioral Scale II, GECEN rating form, and an academic skills rating form (GEVA-SCO), in the records from the MDPH and the school records (ULIS or IME), and dated from within one year before the latest child orientation decision.

SECONDARY OUTCOMES:
Presence of the ID assessment kit results in the records | within one year before the inclusion
  Presence of the results of the neuropsychological tests included in the ID assessment kit: WISC-IV (IQ), Vineland Adaptive Behavioral Scale II, GECEN rating form, and an academic skills rating form (GEVA-SCO), in the records from the MDPH and the school records (ULIS or IME), and dated from within a year before the inclusion in the study.
List of tests available in the children' records, other than the ones from the ID kit. | within one year before the latest child orientation decision
  All the available tests will be listed.
List of tests available in the children's records, other than the ones from the ID kit. | within a year before the inclusion
  All the available tests will be listed
WISC-IV (Wechsler Intelligence Scale for Children 4th edition) | within one year before the latest child orientation decision
  The Intellectual Quotient of the patient will be assessed using a Wechsler scale, adapted to the age of the patient (WISC-IV).
Vineland Adaptive Behavioral Scale II | within one year before the latest child orientation decision
  The Vineland adaptive behavioral scale performed during a semi-structured interview of each child's parents, will allow to assess the adaptive behavior of the child (including communication, daily living skills, socialization, motricity and the global adaptive score).
GECEN rating form (Grille d'Evaluation Comportementale pour Enfants Nisonger | within one year before the latest child orientation decision
  The GECEN rating form (Grille d'Evaluation Comportementale pour Enfants Nisonger) is the French translation of the Nisonger Child Behavior Rating Form and will allow the assessment of behavior disorders including: conduct disorders, anxiety, hyperactivity, automutilation/stereotyped behavior, self-isolation/rituals, sensitivity/susceptibility.
an academic skills rating form | within one year before the latest child orientation decision
  The academic skills rating form will assess 4 domains: the spoken and the written language, the "discovery of the world", and "being a student".
Rehabilitation programs | one year after Day 0
  We will record from the MDPH files the type of rehabilitations that the children had at the latest child orientation decision.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Des PORTES, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No